CLINICAL TRIAL: NCT04000711
Title: Safety and Efficacy of Ambulatory Versus In-hospital Antibiotic Treatment in Pediatric Patients With Cancer and Febrile Neutropenia: a Non-inferiority Multicenter Randomized Clinical Trial
Brief Title: Safety and Efficacy of Ambulatory Versus In-hospital Antibiotic Treatment in Children With Febrile Neutropenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Collaborators: Instituto Nacional de Pediatria (Unknown); Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Martha Josefina Avilés Robles, Chief of Pediatric Infectious Diseases Service, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIM-2014-026; 233555 (Other Grant/Funding Number: Consejo Nacional de Ciencia y Tecnologia (CONACyT) of Mexico)
Record Dates: First submitted 2019-06-24; First posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy-Induced Febrile Neutropenia
Keywords: Fever and neutropenia; Febrile neutropenia; Cancer; Outpatient treatment; Children
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia; Fever; Neutropenia; Febrile Neutropenia; Neoplasms

STUDY DESIGN:
Intervention Model Description: A multicenter, noninferiority randomized clinical trial was conducted in three public hospitals in Mexico City. A complete medical history, physical examination and review of laboratory tests and cultures were performed on all subjects with FN events who were considered low risk. All subjects began receiving intravenous inpatient treatment with cefepime. Subjects were followed-up daily, and those who met the inclusion/exclusion criteria after 48 to 72 hours of in-hospital intravenous treatment were randomly assigned to receive outpatient treatment with oral cefixime or to continue in-hospital intravenous treatment. The treatment was administered by the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient oral antibiotic treatment group. (Experimental): After randomization, participants assigned to receive outpatient treatment with oral cefixime at a dose of 8 mg/kg/day were discharged. Treatment was provided by the researchers. Subjects were evaluated daily at the outpatient clinic of the hospital. All patients underwent a blood count every 48 to 72 hours. FN event resolution was defined as when the patient remained afebrile and the ANC increased to above 500 per microliter. If fever resumed in the outpatient group, they were re-admitted to the hospital to receive intravenous antibiotics. Resolution of the FN event was defined as the end of participation of the subjects in the study, and they were followed up for an additional 72 hours.
  Interventions: Other: Outpatient oral treatment.
- Inpatient intravenous antibiotic treatment group. (Active Comparator): After randomization, participants continued intravenous inpatient antibiotic with cefepime 150 mg/kg/day according to local standard of care guidelines. Subjects were evaluated daily. All patients underwent a blood count every 48 to 72 hours. FN event resolution was defined as when the patient remained afebrile and the ANC increased to above 500 per microliter. If fever resumed, treatment was changed according to clinical guidelines. Resolution of the FN event was defined as the end of participation of the subjects in the study, and they were followed up for an additional 72 hours.
  Interventions: Other: Inpatient intravenous treatment.

INTERVENTIONS:
Other: Outpatient oral treatment. — Participants allocated in oral outpatient group were discharged home with oral antibiotic to continue management. Participants were given Cefixime oral suspension (100 mg/5 mL). Antibiotic was given to the caretakers with written instructions about dosage and time of administration. Dosage indicated was 8 mg/kg/day to be given orally as a single dose (max dose 400 mg/day). Oral antibiotic treatment was given until documented ANC > 500, failure to treatment (restart of fever) or when 14 days of antibiotic were completed (whichever occurred first).
  Arms: Outpatient oral antibiotic treatment group.
Other: Inpatient intravenous treatment. — Participants allocated in the intravenous inpatient group continued receiving Cefepime 150 mg/kg/day every 8 hours (max dose 2 grams per dose or 6 grams per day) according to local standard of care guidelines. Intravenous antibiotic treatment was given until documented ANC > 500, failure to treatment (restart of fever) or when 14 days of antibiotic were completed (whichever occurred first).
  Arms: Inpatient intravenous antibiotic treatment group.

SUMMARY:
Febrile neutropenia (FN) continues to be the infectious complication that most commonly requires hospitalization in pediatric cancer patients undergoing chemotherapy. In recent years, data have been published on the effectiveness of treatment of FN events with oral antibiotics, mainly in developed countries, but data from developing countries continue to be scarce.

Our hypothesis was that early change from initial in-patient intravenous antibiotic treatment to oral outpatient antibiotic treatment in children with cancer and FN is as safe and effective as in-patient intravenous antibiotic management.

The purpose of this clinical study was to determine whether early outpatient oral antibiotic treatment is not inferior in safety and efficacy to in-hospital intravenous antibiotic treatment in pediatric patients with cancer and low-risk FN events.

A multicenter, non-inferiority randomized clinical trial was conducted in three public hospitals in Mexico City. Low-risk FN events were identified in children aged 1 to 18 years. After 48 to 72 hours of receiving intravenous in-hospital antibiotics, children were randomly allocated to receive outpatient oral treatment (cefixime) or to continue in-hospital intravenous treatment (cefepime). Daily monitoring was performed until the resolution of neutropenia. Our outcome of interest was the presence of any unfavorable clinical outcome.

DETAILED DESCRIPTION:
Introduction: Febrile neutropenia (FN) continues to be the infectious complication that most commonly requires hospitalization in pediatric cancer patients undergoing chemotherapy. Classically these patients have been managed as inpatient. In recent years, data have been published on the effectiveness of treatment of FN events with oral antibiotics, mainly in developed countries, but data from developing countries continue to be scarce.

Hypothesis: Our hypothesis was that early change from initial in-patient intravenous antibiotic treatment to oral outpatient antibiotic treatment in children with cancer and FN is as safe and effective as in-patient intravenous antibiotic management.

Objectives: The purpose of this clinical study was to determine whether early outpatient oral antibiotic treatment is not inferior in safety and efficacy to in-hospital intravenous antibiotic treatment in pediatric patients with cancer and low-risk FN events.

Methodology: A multicenter, non-inferiority randomized clinical trial was conducted in three public hospitals in Mexico City. Low-risk FN events were identified in children aged 1 to 18 years.

A complete medical history, physical examination and review of laboratory tests and cultures were performed on all subjects with FN events who were considered low risk. According to local guidelines for the treatment of FN, all subjects began receiving cefepime at a dose of 150 mg/kg/day. Subjects were followed-up daily, and those who met the inclusion/exclusion criteria after 48 to 72 hours of in-hospital intravenous treatment with cefepime were randomly assigned to receive outpatient treatment with oral cefixime at a dose of 8 mg/kg/day or to continue in-hospital intravenous treatment. The treatment was administered by the researchers.

Participants in both treatment groups were evaluated daily by a complete physical examination. Subjects in the outpatient group were evaluated at the outpatient clinic of the hospital. All patients underwent a blood count every 48 to 72 hours. FN event resolution was defined as when the patient remained afebrile and the absolute neutrophil count (ANC) increased to above 500 per microliter. If fever resumed, the antibiotic regimen was modified. If the subjects were in the outpatient group, they were re-admitted to the hospital to receive intravenous antibiotics. Resolution of the FN event was defined as the end of participation of the subjects in the study, and they were followed up for an additional 72 hours.

The occurrence of any of the following conditions was considered an unfavorable clinical outcome: 1) therapeutic failure, defined as the resumption of fever in a patient with persistent neutropenia. For all patients with resumption of fever, the antibiotic regimen was switched, and if the patients were in the outpatient treatment group, they were re-admitted to the hospital; 2) new focus of infection, documented both by the clinical condition and by laboratory and other diagnostic tests; 3) hemodynamic instability, defined as a decrease in blood pressure below the 5th percentile for the patient age that did not revert with the administration of crystalloid solutions; and 4) death.

Sample size: The sample size was calculated to reject a null hypothesis of inferiority, with a non-inferiority margin of presentation of unfavorable clinical outcomes of 15%. A formula including a statistical power of 80% and a one-tailed alpha value of 0.025 was used to calculate the sample size of 2 independent proportions. Based on previous reports of 10% of unfavorable clinical outcomes during the management of FN events, the calculation yielded a total of 63 FN events per group for a total of 126 events.

Randomization: A random sequence balanced by blocks of 4 FN events was generated using a computer program. A physician who did not participate in the subject selection assigned subjects to receive either outpatient oral treatment at home or to continue in-hospital intravenous treatment. If the subjects lived more than 1 hour away from the hospital, they were assigned to a care home to ensure that they could return to the hospital in case of any event. Because the study intervention involved outpatient treatment, the study was open. All patients were provided with the antibiotic free of charge.

Statistical analysis: The focus of analysis was intention-to-treat. For each comparison group, measures of central tendency and dispersion were estimated for continuous variables, and absolute and relative frequencies were determined for discrete and nominal variables. The statistical test performed to test the hypothesis of non-inferiority is very similar to the traditional test for comparison of proportions; the only difference is that the non-inferiority margin is added to the formula, and a p-value < 0.05 confirms non-inferiority. The statistical program STATA version 14.2 was used for the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children from 1 to 18 years of age.
* Underlying cancer diagnosis that presented with fever and neutropenia secondary to chemotherapy and after 48-72 hours of inpatient intravenous treatment with Cefepime, were hemodynamically stable, remained afebrile for at least 24 hours, and did not have a documented source of infection.
* Participants whose caretaker knew how to read and write and accepted to be part of the clinical trial.

Exclusion Criteria:

* Participants with positive cultures.
* Absolute neutrophil count (ANC) < 100/mm3.
* Thrombocytopenia < 30,000/mm3.
* Less than 7 days have passed from the start of the last chemotherapy session.
* Leukemia on remission induction therapy.
* Relapsed leukemia.
* Mucositis grade III or IV.
* Participants with allergy to cefixime.
* Need to receive any other medication intravenously.
* Need of oxygen support, parenteral nutrition or intravenous fluids.
* Oral intolerance.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 117 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-08 (Actual)

PRIMARY OUTCOMES:
Therapeutic failure as unfavorable clinical outcome of children with fever and neutropenia treated with oral outpatient antibiotic. | 17 days after randomization.
  Occurrence of therapeutic failure, defined as the resumption of fever in a patient with persistent neutropenia. For all patients with resumption of fever, the antibiotic regimen was switched, and if the patients were in the outpatient treatment group, they were re-admitted to the hospital.
New focus of infection as unfavorable clinical outcome of children with fever and neutropenia treated with oral outpatient antibiotic. | 17 days after randomization.
  Presence of a new focus of infection, documented both by the clinical condition and by laboratory and other diagnostic tests.
Hemodynamic instability as unfavorable clinical outcome of children with fever and neutropenia treated with oral outpatient antibiotic. | 17 days after randomization.
  Presence of hemodynamic instability, defined as a decrease in blood pressure below the 5th percentile for the patient age that did not revert with the administration of crystalloid solutions.

SECONDARY OUTCOMES:
Presentation of any adverse reaction to any given antibiotic (oral or intravenous) of children with fever and neutropenia treated with oral outpatient vs intravenous inpatient management. | Started on the day of enrollment and concluded 17 days after.
  Moderate and severe adverse reaction to antibiotics given, described as an appreciably harmful or unpleasant reaction, resulting from an intervention related to the use of a medicinal product, which predicts hazard from future administration and warrants prevention or specific treatment, or alteration of the dosage regimen, or withdrawal of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Martha J. Aviles Robles, Principal Investigator — Hospital Infantil de Mexico Federico Gomez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freifeld AG, Bow EJ, Sepkowitz KA, Boeckh MJ, Ito JI, Mullen CA, Raad II, Rolston KV, Young JA, Wingard JR; Infectious Diseases Society of America. Clinical practice guideline for the use of antimicrobial agents in neutropenic patients with cancer: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2011 Feb 15;52(4):e56-93. doi: 10.1093/cid/cir073. PMID 21258094
- [Background] Santolaya ME, Rabagliati R, Bidart T, Paya E, Guzman AM, Morales R, Braun S, Bronfman L, Ferres M, Flores C, Garcia P, Letelier LM, Puga B, Salgado C, Thompson L, Tordecilla J, Zubieta M; Sociedad Chilena de Infectologia; Sociedad Chilena de Hematologia. [Consensus: Rational approach towards the patient with cancer, fever and neutropenia]. Rev Chilena Infectol. 2005;22 Suppl 2:S79-113. Epub 2005 Nov 4. Spanish. PMID 16311689
- [Background] Lehrnbecher T, Phillips R, Alexander S, Alvaro F, Carlesse F, Fisher B, Hakim H, Santolaya M, Castagnola E, Davis BL, Dupuis LL, Gibson F, Groll AH, Gaur A, Gupta A, Kebudi R, Petrilli S, Steinbach WJ, Villarroel M, Zaoutis T, Sung L; International Pediatric Fever and Neutropenia Guideline Panel. Guideline for the management of fever and neutropenia in children with cancer and/or undergoing hematopoietic stem-cell transplantation. J Clin Oncol. 2012 Dec 10;30(35):4427-38. doi: 10.1200/JCO.2012.42.7161. Epub 2012 Sep 17. PMID 22987086
- [Background] Santolaya ME, Alvarez AM, Aviles CL, Becker A, Cofre J, Enriquez N, O'Ryan M, Paya E, Salgado C, Silva P, Tordecilla J, Varas M, Villarroel M, Viviani T, Zubieta M. Prospective evaluation of a model of prediction of invasive bacterial infection risk among children with cancer, fever, and neutropenia. Clin Infect Dis. 2002 Sep 15;35(6):678-83. doi: 10.1086/342064. Epub 2002 Aug 23. PMID 12203164
- [Background] Hakim H, Flynn PM, Srivastava DK, Knapp KM, Li C, Okuma J, Gaur AH. Risk prediction in pediatric cancer patients with fever and neutropenia. Pediatr Infect Dis J. 2010 Jan;29(1):53-9. doi: 10.1097/INF.0b013e3181c3f6f0. PMID 19996816
- [Background] Vidal L, Ben Dor I, Paul M, Eliakim-Raz N, Pokroy E, Soares-Weiser K, Leibovici L. Oral versus intravenous antibiotic treatment for febrile neutropenia in cancer patients. Cochrane Database Syst Rev. 2013 Oct 9;2013(10):CD003992. doi: 10.1002/14651858.CD003992.pub3. PMID 24105485
- [Background] Zapata-Tarrés Marta, Klünder-Klünder Miguel, Cicero-Oneto Carlo, Rivera-Luna Roberto, Ortega-Ríos Velasco Fernando, Cortés Gallo Gabriel et al . Análisis de la atención de las complicaciones durante el tratamiento de niños con leucemia linfoblástica aguda. Bol. Med. Hosp. Infant. Mex.
- [Background] Aviles-Robles M, Ojha RP, Gonzalez M, Ojeda-Diezbarroso K, Dorantes-Acosta E, Jackson BE, Johnson KM, Caniza MA. Bloodstream infections and inpatient length of stay among pediatric cancer patients with febrile neutropenia in Mexico City. Am J Infect Control. 2014 Nov;42(11):1235-7. doi: 10.1016/j.ajic.2014.07.021. Epub 2014 Sep 16. PMID 25234044
- [Derived] Aviles-Robles MJ, Reyes-Lopez A, Otero-Mendoza FJ, Valencia-Garin AU, Penaloza-Gonzalez JG, Rosales-Uribe RE, Munoz-Hernandez O, Garduno-Espinosa J, Juarez-Villegas L, Zapata-Tarres M. Safety and efficacy of step-down to oral outpatient treatment versus inpatient antimicrobial treatment in pediatric cancer patients with febrile neutropenia: A noninferiority multicenter randomized clinical trial. Pediatr Blood Cancer. 2020 Jun;67(6):e28251. doi: 10.1002/pbc.28251. Epub 2020 Mar 20. PMID 32196898